CLINICAL TRIAL: NCT04653194
Title: Efficacy of BIC/F/TAF Versus Standard of Care in the Treatment of New HIV Infection Diagnoses in the Context of 'Test and Treat'
Acronym: BIC-T&T
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chelsea and Westminster NHS Foundation Trust (Other)
Collaborators: Imperial College London (Other); Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRF002; 2019-003208-11 (EudraCT Number)
Record Dates: First submitted 2020-11-27; First posted 2020-12-04 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-01

CONDITIONS: Human Immunodeficiency Virus
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — bictegravir, emtricitabine, tenofovir alafenamide, drug combination; symtuza

STUDY DESIGN:
Intervention Model Description: Open-label 1:1 non-inferiority randomised clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Biktarvy treatment (Experimental): First-line HIV treatment of Biktarvy OD for 48 weeks
  Interventions: Drug: Biktarvy
- Symtuza treatment (Active Comparator): First-line HIV treatment of Symtuza OD for 48 weeks
  Interventions: Drug: Symtuza

INTERVENTIONS:
Drug: Biktarvy — Combination single tablet anti-retroviral therapy: bictegravir 50mg/emtricitabine 200mg/tenofovir alafenamide 25mg
  Arms: Biktarvy treatment
Drug: Symtuza — Combination single tablet anti-retroviral therapy: darunavir 800mg/cobicistat 150mg/emtricitabine 200mg/tenofovir alafenamide 10mg
  Arms: Symtuza treatment

SUMMARY:
The administration of combination antiretroviral therapy (cART) to HIV-infected patients has been associated with a dramatic reduction in AIDS-related morbidity and mortality. Time to cART start is currently approximately 2-4 weeks after diagnosis, mostly deferred for reasons of waiting for baseline blood test results; in particular HIV genotype, CD4 count, OI screen and logistics of a consultant clinical review. Whilst there is a clear rationale for this delay there is a risk of loss to follow-up as well as the potential risk of onward viral transmission. The balance between "readiness" to start ART against pragmatic and practical safe initiation of treatment needs to be tested using currently available safe potent antiretroviral agents in a head-to-head comparison study to allow careful rigorous comparisons of outcomes.

This study will recruit 36 newly diagnosed HIV patients to be started on treatment immediately upon diagnosis. This would optimally be within 7 days, for eligibility to the study up to 14 days will be permissible. Patients will be randomised to one of two open-label combination therapies known to be highly effective; Biktarvy or Symtuza. The patients will receive study treatment for 48 weeks. The two therapies will be compared by the change in HIV viral load from start of treatment to 12 weeks. Further clinical data will be recorded for the trial patients and exploratory investigations undertaken. As those recruited to the trial may not be representative of the full cohort of newly diagnosed HIV patients there will also be data collected on all newly diagnosed patients in a given period. This data will contribute to conclusions on the benefits and issues of implementing test and treat.

DETAILED DESCRIPTION:
There will be an open-label two arm clinical trial with participants randomised to Biktarvy or Symtuza with equal probability. Study treatment will last for 48 weeks.

Baseline - Following confirmatory HIV testing potential participants will have a appointment with a study doctor. Full medical check and medical history undertaken. Patients will be offered opportunity to participate in the study. To avoid unnecessary visits and in line with the study aim of getting patients on treatment rapidly patients can consent on the same day that HIV diagnosis is confirmed to them. Treatment to be initiated following appointment in line with test and treat procedure. Samples will be taken (if not available from previous days) for all initial required tests.

Participants will be given baseline questionnaires that they can return on week 2 visit.

Week 1 call - Call to check drug adherence, adverse events and patient wellbeing.

Week 2 visit - Appointment with study doctor to review all results from initial tests. Following undertaken: viral load; vital signs; adverse events; adherence assessment.

Week 4, 12, 24, 48 Follow-up visits - Full medical review undertaken at each visit including safety blood tests.

Following undertaken: viral load; adverse events; adherence assessment; questionnaires; samples taken for secondary and exploratory objectives. Week 48 visit will be the end of study treatment period.

Follow-up visit - up to 30 days after the week 48 visit there will be a follow-up visit to complete final medical assessment and final adverse events reporting.

Samples will be collected from participants further to those required for stated objectives to be retained for future research into HIV infection.

We will also collect and clinical data cohort of data on all patients newly diagnosed with HIV during a set window.

Clinical data will be collected from their first year after diagnosis.

ELIGIBILITY:
Inclusion Criteria:

1. Is male or female aged 18 years or over.
2. Confirmed diagnosis of HIV-1 as per local clinic definition less than 14 days before day treatment is to be initiated.
3. Is capable of giving informed consent.
4. Is willing to comply with the protocol requirements
5. A female may be eligible to enter and participate in the study if she:

   1. is of non-child-bearing potential defined as either post-menopausal (12 months of spontaneous amenorrhea and ≥ 45 years of age) or physically incapable of becoming pregnant with documented tubal ligation, hysterectomy or bilateral oophorectomy or,
   2. is of child-bearing potential with a negative pregnancy test at Screening (& baseline visit) and agrees to use one of the methods of contraception to avoid pregnancy indicated in Appendix 4 during the study and for a period of 12 weeks after the study.
6. Men who have partners who are women of childbearing potential (WOCBP - definition in Appendix 4) must be using an adequate method of contraception as listed in Appendix 4 to avoid pregnancy in their partner throughout the study and for a period of at least 12 weeks after the study;

Exclusion Criteria:

1. Infected by HIV-2
2. On PEP
3. Use of medications that are know to interact with either treatment B or S
4. Unstable health conditions that according to the opinion of the Investigator suggest the individual should not take part in the trial (including unstable liver diseases, possible opportunistic infections, etc)
5. Women planning pregnancy or who are pregnant or breast feeding. (NB: See section 4.4; Withdrawal Criteria and Section 10.4; Collection and Follow up of Adverse Events if pregnancy does occur in a trial subject)
6. Ongoing malignancy other than cutaneous Kaposi's sarcoma, basal cell carcinoma, or resected, non-invasive cutaneous squamous cell carcinoma, or cervical intraepithelial neoplasia; other localized malignancies require agreement between the investigator and the Study medical monitor for inclusion of the subject prior to randomisation.
7. Known acute or chronic viral hepatitis including, but not limited to, A, B, or C
8. Any investigational drug within 30 days prior to the trial drug administration
9. Any other condition (including illicit drug use or alcohol abuse) or laboratory results which, in the investigator's opinion, interfere with assessments or completion of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2020-09-30 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Rate of HIV viral load response to first-line anti-retroviral treatment | Baseline to 12 weeks
  Change from baseline to week 12 in log10 HIV RNA level recorded in viral load assays.

SECONDARY OUTCOMES:
Absolute efficacy in achieving viral suppression of newly diagnosed HIV infection. | 2 weeks, 4 weeks, 12 weeks, 24 weeks, 48 weeks
  Proportion of participants achieving viral suppression at study visits as defined both by HIV copies < 20/ml and HIV copies < 50 ml
Adverse events occurrence | Baseline to 48 weeks
  Frequency and severity of occurrence of adverse events in study participants
Viral resistance occurrence | Baseline to 48 weeks
  Frequency of occurrence of confirmed viral resistance to study interventions

CONTACTS AND LOCATIONS:
Overall Officials: Marta Boffito, MD PhD FRCP, Principal Investigator — Chelsea and Westminster NHS Foundation Trust
Locations (3):
- United Kingdom (3):
  - Brighton and Sussex University Hospitals NHS Trust Lawson Unit Royal Sussex County Hospital, Brighton
  - Chelsea and Westminster Hospital NHS Foundation Trust, London
  - Imperial College Healthcare NHS Trust, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Khawaja AA, Whitlock G, Fidler S, Soler-Carracedo A, Henderson M, Taylor GP, Boffito M, Emerson M. Evaluation of the effect of 48 weeks of BIC/F/TAF and DRV/c/F/TAF on platelet function in the context of rapid ART start. HIV Res Clin Pract. 2025 Dec;26(1):2447015. doi: 10.1080/25787489.2024.2447015. Epub 2025 Jan 7. PMID 39763430